CLINICAL TRIAL: NCT03620825
Title: The Effect of Dehydration on Intestinal Permeability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Örebro University, Sweden (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2017/463
Record Dates: First submitted 2018-07-30; First posted 2018-08-08 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Dehydration; Indomethacin
MeSH Terms: conditions — Dehydration | interventions — Indomethacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dehydration by sauna exposure (Experimental): Participants dehydrate using sauna exposure until they lose 3% of their body weight.
  Interventions: Other: Dehydration by sauna exposure
- Indomethacin - Positive control (Active Comparator): Indomethacin is administered to induce increased intestinal permeability
  Interventions: Drug: Indomethacin
- Negative control (No Intervention): No intervention is performed

INTERVENTIONS:
Other: Dehydration by sauna exposure — Participants repeatedly undergo sauna exposures until they loose 3% of their body weight.
  Arms: Dehydration by sauna exposure
Drug: Indomethacin — Participants take indomethacin in tablet form the evening before and the morning of the visit to induce intestinal permeability
  Arms: Indomethacin - Positive control

SUMMARY:
In this study, the effect of dehydration by sauna exposure on the intestinal permeability in 20 healthy subjects is investigated. Participants attend three visits: 1) Sauna visit (to achieve 3% dehydration), 2) Positive control visit (intake of indomethacin which is known to increase intestinal permeability), 3) Negative control visit. At all visits, saliva samples, blood samples, faecal samples, saliva samples are collected and the multi-sugar permeability test is performed. In this test, participants drink a sugar solution and then urine collect urine for 5 and 24 h. The ratio of the sugars detected in the urine by liquid chromatography/mass spectometry is a reflection of the intestinal permeability. Saliva samples are collected for assessment of cortisol, a stress marker. Blood and faecal samples are collected for assessment of markers of intestinal barrier function and inflammation.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent prior to any study related procedures
2. Age > 18 till <50
3. Willing to abstain from probiotic products or medications known to alter gastrointestinal function throughout the study

Exclusion Criteria:

1. Abdominal surgery which might influence gastrointestinal function, except appendectomy and cholecystectomy.
2. Current diagnosis of hypertension.
3. Current diagnosis of psychiatric disease.
4. Over 100kg or with a BMI over 35.
5. Systemic use of steroids in the last 6 weeks.
6. Use of antibiotics or antimicrobial medication in the last month.
7. Daily usage of nonsteroidal anti-inflammatory drugs in the last 2 months or incidental use in the last 2 weeks prior to screening.
8. Usage of medications that could affect the barrier function, except oral contraceptives, during the 14 days prior to screening.
9. Diagnosed inflammatory gastrointestinal disease.
10. Known organic gastrointestinal disease (e.g. irritable bowel syndrome, inflammatory bowel disease, chronic diarrhoea or constipation).
11. History of or present gastrointestinal malignancy or polyposis.
12. Recent (gastrointestinal) infection (within last 6 months).
13. Eosinophilic disorders of the gastrointestinal tract.
14. Current communicable disease (e.g. upper respiratory tract infection).
15. Malignant disease and /or patients who are receiving systemic anti-neoplastic agents).
16. Chronic neurological/neurodegenerative diseases (e.g. Parkinson's disease, multiple sclerosis).
17. Autoimmune disease and/or patients receiving immunosuppressive medications.
18. Major relevant allergies (e.g. food allergy, multiple allergies).
19. Chronic pain syndromes (e.g. fibromyalgia)
20. Chronic fatigue syndrome
21. Regular use of probiotics in the last 6 weeks.
22. Smoking and/or chewable tobacco.
23. Planned changes to current diet or exercise regime.
24. Use of laxatives, anti-diarrhetics, anti-cholinergics within last 4 weeks prior to screening.
25. Use of immunosuppressant drugs within last 4 weeks prior to screening.
26. Women: Pregnancy, lactation.
27. Abuse of alcohol or drugs.
28. Any disease/condition which in the investigator's opinion could interfere with the intestinal barrier function.
29. Any clinically significant disease/condition which in the investigator's opinion could interfere with the results of the trial.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-03-17 (Actual); Primary Completion 2018-06-21 (Actual); Study Completion 2018-06-21 (Actual)

PRIMARY OUTCOMES:
Change in small intestinal permeability measured as the urinary lactulose/rhamnose secretion ratio compared to negative control | 1-2 weeks

SECONDARY OUTCOMES:
Change in whole gut permeability measured as the urinary sucralose/erythritol secretion ratio compared to negative control | 1-2 weeks
Change in colonic permeability measured as the urinary sucralose/erythritol secretion ratio compared to negative control | 1-2 weeks
Change in gastroduodenal permeability measured as urinary sucrose excretion | 1-2 weeks
Change in quantity of intestinal permeability markers in blood | 1-2 weeks
  e.g. fatty acid binding proteins
Change in salivary cortisol levels | 1-2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Brummer, MD, PhD, Principal Investigator — Örebro University, Sweden
Locations (1):
- Örebro University, Örebro, Örebro County, Sweden

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared

REFERENCES:
- [Derived] Roca Rubio MF, Eriksson U, Brummer RJ, Konig J. Sauna dehydration as a new physiological challenge model for intestinal barrier function. Sci Rep. 2021 Jul 30;11(1):15514. doi: 10.1038/s41598-021-94814-0. PMID 34330970